CLINICAL TRIAL: NCT04747600
Title: Outcomes of Surgical Resection of Pancreatic Cystic Neoplasms Based on the European Expert Consensus Statement: A Prospective Observational Study.
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, assistant professour of general and laparoscopic surgery, Zagazig University
Other Study IDs: zagazig PCN
Record Dates: First submitted 2021-02-07; First posted 2021-02-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- serous cystic neoplasms
  Interventions: Procedure: surgical resection
- mucinous cystic neoplasms
  Interventions: Procedure: surgical resection
- intra-papillary mucinous neoplasms
  Interventions: Procedure: surgical resection
- solid pseudo-papillary neoplasms
  Interventions: Procedure: surgical resection

INTERVENTIONS:
Procedure: surgical resection — surgical resection

SUMMARY:
Introduction: Pancreatic cystic neoplasms (PCNs) comprise neoplasms with a wide range of benign and malignant varieties. The most common include serous cystic neoplasms (SCNs), mucinous cystic neoplasms (MCNs), intraductal papillary mucinous neoplasms (IPMNs), and solid pseudo-papillary neoplasms (SPPNs).

Endoscopic ultrasonography (EUS), computed tomography (CT) and magnetic resonance (MR) are used to diagnose different PCNs types. The cyst fluid aspiration and analysis is performed in difficult differential diagnosis. Frequently, amylase and CEA levels are measured. The choice of surgery depends on cyst location and size and includes pancreatico-duodenectomy or distal pancreatectomy.

Objectives: The aim of this study was to evaluate the outcomes after pancreatic surgery when adopted as the management of true exocrine epithelial cystic neoplasms.

DETAILED DESCRIPTION:
Introduction: Pancreatic cystic neoplasms (PCNs) comprise neoplasms with a wide range of benign and malignant varieties. The most common include serous cystic neoplasms (SCNs), mucinous cystic neoplasms (MCNs), intraductal papillary mucinous neoplasms (IPMNs), and solid pseudo-papillary neoplasms (SPPNs).

Endoscopic ultrasonography (EUS), computed tomography (CT) and magnetic resonance (MR) are used to diagnose different PCNs types. The cyst fluid aspiration and analysis is performed in difficult differential diagnosis. Frequently, amylase and CEA levels are measured. The choice of surgery depends on cyst location and size and includes pancreatico-duodenectomy or distal pancreatectomy.

Objectives: The aim of this study was to evaluate the outcomes after pancreatic surgery when adopted as the management of true exocrine epithelial cystic neoplasms.

Patients and methods: Between June 2014 and January 2018, 63 patients referred to our tertiary referral center with diagnosis of true exocrine cystic neoplasms of the pancreas accepted for surgery were included in the present prospective cohort study. Patients were categorized according to preoperative diagnosis into: serous cystic neoplasms (Group A: 30 patients), mucinous cystic neoplasms (Group B: 13 patients), intra-papillary mucinous neoplasms (Group C: 9 patients), whereas the last 5 patients diagnosed as solid pseudo-papillary neoplasms (Group D). Demographic data, perioperative data and univariate analysis for malignancy, recurrence and pancreatic fistula were collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* any Age
* both sex,
* expected R0 resection,
* Tumor of any size,
* no previous pancreatic surgery with diagnosis of True exocrine pancreatic cystic neoplasms

Exclusion Criteria:

* endocrinal pancreatic tumors,
* solid pancreatic tumors,
* previous pancreatic surgery,
* recurrent pancreatic tumor,
* Combined operation,
* prior history of any malignancy and misdiagnosed cases discovered on postoperative pathological cases as pancreatic pseudo-cyst or endocrine tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 63 patients with a clinical diagnosis of true exocrine pancreatic cystic neoplasms were enrolled in this prospective cohort study as a comprehensive sampling in our hepato-biliary pancreatic unit of our university hospital between June 2014 to January 2018. They were categorized into 4 groups: Group A(30 patients)that were diagnosed as serous cystic neoplasms, Group B(19 patients) that were diagnosed as mucinous cystic neoplasms, Group C(9 patients )that were diagnosed as intra-ductal papillary mucinous neoplasms and Group D(5 patients ) that were diagnosed as solid pseudo-papillary neoplasms.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
the incidence of the pancreatic fistula | 30 days postoperatively
  detect pancreatic fistula by concentration of amylase level in drain

SECONDARY OUTCOMES:
recurrence rate in percentage | 2.5 years
  rate of recurrence after resection by computed tomography

IPD SHARING:
Plan to Share IPD: Undecided